CLINICAL TRIAL: NCT07097623
Title: Optimal Acute Adult Psychiatric In-patient Care in Hong Kong: a Mixed-method Study
Brief Title: Optimal Acute Adult Psychiatric In-patient Care in Hong Kong
Status: Not yet recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Nethersole Institute of Continuing Holistic Health Education (NICHE) (Unknown)
Responsible Party: Principal Investigator, Dennis Chak Fai Ma, Assistant Professor of Practice, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20231025005
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Hospitalization
Keywords: adult psychiatric inpatient care, optimal bed number

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Psychiatric nurses
  Interventions: Other: respond to 3 rounds of online Delphi surveys
- Service users
  Interventions: Other: attend an individual semi-structured interview
- Family caregivers
  Interventions: Other: attend an individual semi-structured interview

INTERVENTIONS:
Other: respond to 3 rounds of online Delphi surveys — In the first round, the responses of the participants will be collected, coded, and categorised into several themes/factors anonymously. In the second round, the participants will obtain the controlled feedback of all other participants and rate the level of agreement of the factors using a 5-point Likert scale ('strongly agree', 'agree', 'neither agree or disagree', 'disagree', and 'strongly disagree'; or 'essential', 'important', 'don't know/depends', 'unimportant', and 'should not be considered'). In the third round, the participants will rank the importance of the factors. In each round, the participants will be expected to complete the survey within one month.
  Groups: Psychiatric nurses
Other: attend an individual semi-structured interview — The individual semi-structured interview will be audio-recorded, last for 45 minutes at maximum, and carried out by a trained and independent research assistant in a meeting room of PolyU or a room affiliated with the respective acute wards of the participating hospitals.
  Groups: Family caregivers; Service users

SUMMARY:
This mixed-method study aims to evaluate the optimal number of hospital beds and quality of acute adult psychiatric inpatient care in Hong Kong using online Delphi surveys for psychiatric nurses and individual interviews for service users with mental health conditions and family caregivers. The main question it aims to answer is:

What are the consensus points for quality acute adult psychiatric inpatient care in Hong Kong from psychiatric nurses, service users, and caregivers?

Psychiatric nurses will respond to three rounds of online Delphi surveys, while service users and caregivers will attend individual semi-structured interviews.

DETAILED DESCRIPTION:
The deinstitutionalisation movement has been implemented since the 1950s, particularly in the UK and the US. Evidence of psychiatric community care has been well-documented, showing improvements in quality of life, increased autonomy, a reduction in psychiatric readmissions, and a shorter length of hospitalisation. However, this movement has not been universally adopted, and a few drawbacks have emerged in the past decade. Increased social risk aversion, such as homicides and a higher incidence of comorbidity of severe mental illnesses and substance abuse, has led to a growing demand for psychiatric inpatient services. Additionally, insufficient long-term community residential care was associated with untreated service users living in prisons or experiencing homelessness. The reduction in psychiatric beds was also associated with an increased prison population in the UK, Central and Eastern Europe, Central Asia, and South America.

From 2000 to 2014, 55% of 161 nations had stable or increasing levels of institutionalisation (> 1% annually). Several national characteristics, for example, population density and the percentage of the population living in urban areas, were negatively associated with deinstitutionalisation. The findings argued that the development of deinstitutionalisation should carefully consider the maturity of local psychiatric facilities and systems; otherwise, achieving a balance of optimal psychiatric inpatient care and deinstitutionalisation may be difficult. This imbalance can lead to a shift of service users into the criminal justice system. Moreover, deinstitutionalisation was positively associated with acute admission rates and bed occupancy. A viewpoint published in JAMA discussed the dilemma of psychiatric inpatient care versus community psychiatric development in the US, calling for integrated, patient-centred long-term psychiatric hospital and outpatient care for individuals with chronic, serious mental health conditions.

Since 2010, the Hong Kong government has made extensive efforts and committed significant resources to community psychiatric care, including the extended hospital community psychiatric services (CPS) and district-based community mental health centres. However, these initiatives led to a reduction in emergency psychiatric admissions, which is one of the key quality indicators of community mental health care, for neuroses, but not for other diagnoses of mental health conditions, particularly for severe mental illnesses. A balanced mental health system that integrates psychiatric inpatient and CPS care, especially for severe mental illnesses with notable risks of violence and suicide, should be actively reconsidered. As psychiatric inpatient service capacity decreases during active deinstitutionalisation, optimal psychiatric inpatient care has often been overlooked, which may hinder the development of specialised inpatient services and pose risks to clinical quality and safety due to overcrowded ward environments and increased admission turnover rates, commonly known as the 'revolving door' effect.

ELIGIBILITY:
I. Psychiatric nurses

Inclusion Criteria:

* working in the Hospital Authority on a full-time basis,
* with ≥ 10 years post-registration experience, and
* able to read and understand English

Exclusion Criteria:

* without working experience in adult psychiatry

II. Service users

Inclusion Criteria:

* aged 18-64
* able to read and communicate in Cantonese, and
* being discharged within a year

Exclusion Criteria:

* having a co-morbidity of learning disability, organic/neurological conditions, or substance misuse disorder

III. Family caregivers

Inclusion Criteria:

* aged 18 or above, and
* able to read and communicate in Cantonese

Exclusion Criteria:

* having active psychiatric conditions

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Participants will be recruited from the psychiatric departments within four clinical clusters of the Hong Kong Hospital Authority.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
consensus on the optimal number and minimum number of psychiatric inpatient beds as assessed using two numeric questions in the Delphi survey | 3-6 months
  To reach an expert consensus, ≥ 85% of numeric responses fall within the first and third quartiles of the responses
consensus on the optimal nurse-patient ratio as assessed using a numeric question in the Delphi survey | 3-6 months
  To reach an expert consensus, ≥ 85% of numeric responses fall within the first and third quartiles of the responses
consensus on the optimal length of stay by diagnoses as assessed using a numeric question in the Delphi survey | 3-6 months
  To reach an expert consensus, ≥ 85% of numeric responses fall within the first and third quartiles of the responses
consensus on factors contributing to the optimal numbers of psychiatric inpatient beds as assessed using four open-ended questions in the Delphi survey | 3-6 months
  To reach an expert consensus, ≥ 85% agreement with the two favourable responses (e.g., 'strongly agree' and 'agree') on items is achieved
consensus on recommendations for achieving optimal acute adult psychiatric inpatient services as assessed using five open-ended questions in the Delphi survey | 3-6 months
  To reach an expert consensus, ≥ 85% agreement with the two favourable responses (e.g., 'strongly agree' and 'agree') on items is achieved
experience and expectation of optimal adult psychiatric inpatient care as assessed using individual interviews | 1-3 months
  certain themes will be generated by thematic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chak Fai Ma, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University